CLINICAL TRIAL: NCT01203098
Title: A Phase 2b, Randomized, Multi-Dose Efficacy,Safety Study of the Oral Factor Xa Inhibitor DU-176b Versus Enoxaparin Sodium for Prevention of Venous Thromboembolism in Patients After Total Hip Arthroplasty (STARS J-2)
Brief Title: A Phase 2b Study of DU-176b, Prevention of Venous Thromboembolism in Patients After Total Hip Arthroplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DU176b-B-J209
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Results first posted 2015-02-09 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2015-02

CONDITIONS: Venous Thromboembolism; Thromboembolism; Thrombosis; Embolism and Thrombosis; Deep Vein Thrombosis; Arthroplasty, Replacement, Hip
Keywords: prevention; venous thromboembolism; edoxaban; anticoagulants
MeSH Terms: conditions — Venous Thromboembolism; Thromboembolism; Thrombosis; Embolism and Thrombosis; Venous Thrombosis | interventions — edoxaban; enoxaparin sodium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DU-176b 30mg once daily (Experimental): DU-176b 30 mg tablets, oral once daily for 2 weeks initiated within 6 to 24 hours after surgery
  Interventions: Drug: DU-176b 30mg
- Enoxaparin sodium twice daily (Active Comparator): Enoxaparin sodium 20mg (=2000IU) / 0.2mL twice daily, subcutaneous injection for 2 weeks, initiated within 24 to 36 hours after surgery
  Interventions: Drug: Enoxaparin sodium 20 mg (=2000IU)
- DU-176b 15mg once daily (Experimental): DU-176b 15mg tablets, oral once daily for 2 weeks initiated within 6 to 24 hours after surgery
  Interventions: Drug: DU-176b 15mg

INTERVENTIONS:
Drug: DU-176b 15mg — DU-176b 15 mg tablets oral, once daily for 2 weeks initiated within 6 to 24 hours after surgery.
  Other Names: edoxaban
  Arms: DU-176b 15mg once daily
Drug: DU-176b 30mg — DU-176b 30 mg tablets, oral once daily for 2 weeks initiated within 6 to 24 hours after surgery.
  Other Names: edoxaban
  Arms: DU-176b 30mg once daily
Drug: Enoxaparin sodium 20 mg (=2000IU) — Enoxaparin sodium 20 mg (=2000IU) / 0.2ml twice daily, subcutaneous injection for 2 weeks initiated within 24 to 36 hours after surgery.
  Arms: Enoxaparin sodium twice daily

SUMMARY:
The objective of this study is to compare the efficacy, safety of DU-176b 30mg or DU-176b 15mg versus enoxaparin sodium for the prevention of venous thromboembolism in patients after elective total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing unilateral total hip arthroplasty
2. Patients who are 20-84 years olds

Exclusion Criteria:

1. Subjects with risks of hemorrhage
2. Subjects with thromboembolic risks
3. Subjects who weigh less than 40 kg
4. Subjects who are pregnant or suspect pregnancy, or subjects who want to become pregnant

Ages: 20 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2008-07; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Fuji, Principal Investigator — Osaka Koseinenkin Hospital
Locations (3):
- Japan (2):
  - Osaka
  - Tokyo
- Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Fuji T, Wang CJ, Fujita S, Kawai Y, Kimura T, Tachibana S. Safety and efficacy of edoxaban, an oral factor xa inhibitor, for thromboprophylaxis after total hip arthroplasty in Japan and Taiwan. J Arthroplasty. 2014 Dec;29(12):2439-46. doi: 10.1016/j.arth.2014.05.029. Epub 2014 Jun 9. PMID 25047458

RESULTS

PARTICIPANT FLOW:
Groups:
- DU-176b 15 mg: DU-176b 15 mg tablets, oral once daily for 2 weeks
- DU-176b 30 mg: DU-176b 30 mg tablets oral, once daily for 2 weeks
- Enoxaparin Sodium 20mg (2000IU): Enoxaparin sodium 20 mg (=2000IU) / 0.2ml twice daily, subcutaneous injection for 2 weeks
Period: Overall Study
Arm/Group | DU-176b 15 mg | DU-176b 30 mg | Enoxaparin Sodium 20mg (2000IU)
Started | 89 | 86 | 89
Safety Analysis Dataset | 89 | 85 | 87
Completed | 83 | 82 | 78
Not Completed | 6 | 4 | 11
Not completed — Adverse Event | 3 | 1 | 7
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Physician Decision | 2 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Number of baseline participants reflects the efficacy analysis population
Groups:
- Total: Total of all reporting groups
Arm/Group | DU-176b 15 mg | DU-176b 30 mg | Enoxaparin Sodium 20mg (2000IU) | Total
Number analyzed (Participants) | 78 | 72 | 74 | 224
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (10.3) | 60.6 (9.6) | 58.9 (10.7) | 60.3 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 69 | 59 | 191
  Male | 15 | 3 | 15 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 78 | 72 | 74 | 224
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 3 | 2 | 4 | 9
  Japan | 75 | 70 | 70 | 215

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Venous Thromboembolism Events
Description: The primary efficacy endpoint was the proportion of subjects who experienced at least one of the thromboembolic events listed below during the period from the start of study treatment to the venography at the end of study treatment.
  * Lower extremity DVT confirmed by bilateral venography at the end of study treatment
  * Definite diagnosis of symptomatic PE
  * Symptomatic DVT confirmed before the venography at the end of study treatment The objectives were to verify the non-inferiority of edoxaban to enoxaparin with regard to prevention of VTE
Time Frame: 2 weeks
Population: The FAS was defined as all subjects enrolled in the study, but excluded those who had significant GCP violations, who had not received any doses of the study drug, or those who did not develop symptomatic DVT or PE, but in whom venography was not appropriately performed.
Measure: Number (95% Confidence Interval); unit: percent of participants with VTE event
Arm/Group | DU-176b 15 mg | DU-176b 30 mg | Enoxaparin Sodium 20mg (2000IU)
Number analyzed (Participants) | 78 | 72 | 74
percent of participants with VTE event | 3.8 [0.0 to 8.1] | 2.8 [0.0 to 6.6] | 4.1 [0.0 to 8.5]
Statistical Analysis 1: Comparison: DU-176b 30 mg vs Enoxaparin Sodium 20mg (2000IU); Primary analyses were performed on proportion of subjects who experienced thromboembolic events defined as primary efficacy endpoint (incidence of thromboembolic events); incidence of thromboembolic events and its 95% confidence interval (CI) were calculated by treatment group, and difference between DU-176b 15 mg and 30 mg groups and its 95% CI were also calculated. For reference, difference between enoxaparin group and each DU-176b group and its 95% CI of each were calculated; Test type: Superiority or Other; Cox Proportional Hazard = -1.3, 95% CI 2-sided [-7.2 to 4.6]
Statistical Analysis 2: Comparison: DU-176b 15 mg vs DU-176b 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Cox Proportional Hazard = 1.1, 95% CI 2-sided [-4.6 to 6.8]

2. Secondary Outcome: Incidence of Major Bleeding or Clinically Relevant Non-major Bleedings.
Time Frame: 2 weeks
Population: The Safety Analysis Set was defined as all subjects who were enrolled in the study, but excluded those who had significant GCP violations, who did not receive any doses of the study drug, or who had no safety data after the start of study treatment
Measure: Number (95% Confidence Interval); unit: percentage of subjects with bleeds
Arm/Group | DU-176b 15 mg | DU-176b 30 mg | Enoxaparin Sodium 20mg (2000IU)
Number analyzed (Participants) | 89 | 85 | 87
percentage of subjects with bleeds | 2.2 [0.3 to 7.9] | 1.2 [0.0 to 6.4] | 2.3 [0.3 to 8.1]

ADVERSE EVENTS:
Description: The Safety Analysis Set was defined as all subjects who were enrolled in the study, but excluded those who had significant GCP violations, who did not receive any doses of the study drug, or who had no safety data after the start of study treatment
Arm/Group | DU-176b 15 mg | DU-176b 30 mg | Enoxaparin Sodium 20mg (2000IU)
Serious Adverse Events (participants affected / at risk) | 1/89 | 2/85 | 1/87
Other Adverse Events (participants affected / at risk) | 58/89 | 60/85 | 72/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DU-176b 15 mg (N=89) | DU-176b 30 mg (N=85) | Enoxaparin Sodium 20mg (2000IU) (N=87)
dislocation of joint prothesis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
vertigo positional (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DU-176b 15 mg (N=89) | DU-176b 30 mg (N=85) | Enoxaparin Sodium 20mg (2000IU) (N=87)
nasopharyngitis (Infections and infestations) | 5 (5) | 5 (5) | 3 (3)
diarrhea (Gastrointestinal disorders) | 7 (7) | 5 (5) | 6 (6)
haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 6 (7)
alanine aminotransferase increased (Investigations) | 18 (18) | 8 (8) | 36 (36)
aspartate aminotransferase increased (Investigations) | 7 (7) | 3 (3) | 25 (25)
gamma glutamyltransferase (Investigations) | 11 (11) | 14 (14) | 26 (26)
blood urine present (Investigations) | 8 (8) | 7 (9) | 6 (6)
blood alkaline phosphatase increased (Investigations) | 2 (2) | 3 (3) | 9 (9)
dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 4 (5)
headache (Nervous system disorders) | 4 (4) | 2 (2) | 5 (5)
dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 4 (5)
eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 4 (4)
pruritis (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3) | 3 (3)
blood triglycerides increased (Investigations) | 1 (1) | 0 (0) | 4 (4)
abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
stomach discomfort (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3)
vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2)
rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 2 (2)
skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1)
blood lactate dehydrogenase increased (Investigations) | 2 (2) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall not publish the results of the Study at any time without the prior written approval of Sponsor.